CLINICAL TRIAL: NCT02117037
Title: Prognostic Value of Biomarkers Associated With Endothelial Progenitor Cells Mobilization in Acute Coronary Syndromes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-04
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Acute Coronary Syndromes
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study of PEC markers and chemokines/ chemokine recep (Other): blood sample for dosage and study of PEC markers and chemokines/ chemokine receptors
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample

SUMMARY:
This prospective study aimed to validate a new prognostic approach of endothelial progenitor cells associated biomarkers in patients with acute coronary syndromes . Recruitment is made prospectively by two centers of Inter -region South Mediterranean,

ELIGIBILITY:
Inclusion Criteria:

* acute coronary syndrome (ST + < 12 hours and ST- high risk or intermediate risk ),which there is an indication of percutaneous coronary intervention.

Exclusion Criteria:

* Cancer
* Chronic inflammatory disease
* Infectious disease
* Erythrocyte <4 G/l
* Thrombopénia less than 100 000/mm3 ;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
evaluate the value of circulating endothelial progenitor cells quantification in the initial phase of ACS in predicting the occurrence of a major cardiovascular event (ECVM ) at 1 year. | one year

SECONDARY OUTCOMES:
determine the technical characteristics (sensitivity and specificity) and predictive value of the number of PEC | one day , one month , one year

OTHER OUTCOMES:
determine the technical characteristics (sensitivity and specificity) and performance (technical and predictive) of chemokines / receptors expression in the occurrence of ECVM | one day, one month ,one year
Determine the above performance in the subgroup of patients defined as incompletely revascularized (at least a residual stenosis < 70%) | one year

CONTACTS AND LOCATIONS:
Locations (1):
- assistance Publique Hopitaux de Marseille, Marseille, France